CLINICAL TRIAL: NCT03755154
Title: Phase I, Open Label, Non-randomised, Non-comparative, Multi-center Study, Evaluating S65487, a Bcl-2 Inhibitor Intravenously Administered, in Patients With Relapsed or Refractory Acute Myeloid Leukemia, Non Hodgkin Lymphoma, Multiple Myeloma or Chronic Lymphocytic Leukemia
Brief Title: Study of a New Intravenous Drug, Called S65487, in Patients With Acute Myeloid Leukemia, Non Hodgkin Lymphoma, Multiple Myeloma or Chronic Lymphocytic Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was prematurely terminated on 14th March 2023 for strategic considerations due to the limited efficacy seen with this treatment in monotherapy. This decision was not based on any safety concerns.
Sponsor: Institut de Recherches Internationales Servier (Other)
Collaborators: ADIR, a Servier Group company (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL1-65487-002; 2018-004170-97 (EudraCT Number)
Record Dates: First submitted 2018-11-13; First posted 2018-11-27 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Relapsed or Refractory Acute Myeloid Leukemia; Relapsed or Refractory Non-Hodgkin Lymphoma; Relapsed or Refractory Multiple Myeloma; Relapsed or Refractory Chronic Lymphocytic Leukemia
Keywords: Leukemia; Lymphoma; Myeloma; Dose-escalation
MeSH Terms: conditions — Recurrence; Leukemia, Myeloid, Acute; Lymphoma, Non-Hodgkin; Multiple Myeloma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia; Lymphoma; Neoplasms, Plasma Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- S65487 - initial scheme (Experimental)
  Interventions: Drug: S65487- initial scheme
- S65487 - alternative scheme (Experimental)
  Interventions: Drug: S65487 - alternative scheme

INTERVENTIONS:
Drug: S65487- initial scheme — S65487 is administered as single agent via i.v. infusion once a week on a 3-week cycle.
  Arms: S65487 - initial scheme
Drug: S65487 - alternative scheme — S65487 is administered in 3 to 5 i.v. infusions the first week of each cycle then once a week on the rest of the 3-week cycle.
  Arms: S65487 - alternative scheme

SUMMARY:
The purpose of this first in human study is to assess safety, tolerability, Pharmacokinetic (PK) and preliminary clinical activity and to estimate the Maximum Tolerated Doses (MTD(s))/ Recommended Phase 2 Doses (RP2D(s)) of S65487 as single agent administered intravenously (i.v.) in adult patients with refractory or relapsed Acute Myeloid Leukemia (AML), Non-Hodgkin Lymphoma (NHL), Multiple Myeloma (MM) or Chronic Lymphocytic Leukemia (CLL).

DETAILED DESCRIPTION:
This study is designed in two parts: one part for dose escalation, one part for dose expansion.The dose escalation part will be followed by expansion part at the MTD(s)/RP2D(s)

This study will utilize an adaptative Bayesian Logistic Regression model to guide dose escalation and estimate the MTD(s) based on the Dose Limiting Toxicity (DLT) relationship(s) for S65487 in the indications.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cytologically confirmed and documented de novo, secondary or therapy-related AML, excluding acute promyelocytic leukaemia with relapsed or refractory disease without established alternative therapy. Or patients with measurable confirmed Multiple Myeloma (IMWG) with relapsed or refractory disease who have previously received at least three lines of treatment and without established alternative therapy. Or patients with histologically and measurable confirmed Non Hodgkin Lymphoma defined as Diffuse Large B cell Lymphoma (DLBCL), Follicular Lymphoma (FL), Mantle Cell Lymphoma (MCL), Marginal Zone Lymphoma (MZL), High-Grade B cell Lymphoma with relapsed or refractory disease who have received at least two lines of therapy (including rituximab) and without established alternative therapy. Or patients with Chronic Lymphocytic Leukemia (CLL) who have relapsed or are refractory (except treatment failure), as defined per iwCLL, from venetoclax treatment and without established alternative therapy.
* ECOG (Eastern Cooperative Oncology Group) performance status ≤ 2.
* For NHL, MM patients and CLL patients: haematological function (independent of any growth factor support) based on the last assessment performed before inclusion, defined as: absolute neutrophil count (ANC) ≥ 1 x 109/L, haemoglobin ≥ 8 g/dL, platelet count ≥ 50 x 109/L for NHL and MM patients, platelet count ≥ 30 x 109/L for CLL patients.
* For AML patients: circulating Blood White Cell count (WBC count) < 25 x 109/L (with or without use of hydroxycarbamide/leukapheresis) based on the last assessment performed before inclusion.
* Adequate renal function based on the last assessment performed before inclusion, assessed as Glomerular Filtration Rate (GFR) using Modification of Diet in Renal Disease (MDRD) Formula.
* Adequate hepatic function based on the last assessment performed before inclusion.

Exclusion Criteria:

* Pregnancy, breastfeeding or possibility of becoming pregnant during the study.
* Participation in another interventional study at the same time or another interventional study requiring investigational treatment intake within 3 weeks or at least 5 half-lives (whichever is longer) prior to the first S65487 administration.
* Participant already enrolled in the study (informed consent signed) and has received at least one dose of S65487.
* Patients who have not recovered from toxicity of previous anticancer therapy, including grade ≥ 2 non-hematologic toxicity, prior to the first IMP administration (including peripheral neurotoxicity). Certain toxicities will not be considered in this category (e.g. alopecia).
* Patients refractory to a previous treatment with a Bcl-2 inhibitor.
* For AML patients : Allogenic stem cell transplant within 3 months before the first IMP administration and/or patients who still receive immunosuppressive treatment within 3 months before the first IMP administration and/or patients with active Graft-versus-host disease within 3 months before the first IMP administration and/or patient who receive donor lymphocyte infusion (DLI) within 3 months before the first IMP administration.
* For NHL, MM and CLL patients : Prior allogenic stem cell transplant before the first IMP administration and/or Autologous stem cell transplant within 3 months before the first IMP administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2023-11-06 (Actual); Study Completion 2023-11-06 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicity (DLT) | until the end of the first cycle (each cycle is 21days)
  Safety criterion
Incidence and severity of Adverse Events | through study completion an average of 6 months
  Safety and tolerability criteria
Incidence and severity of Serious Adverse Events | through study completion an average of 6 months
  Safety and tolerability criteria
Number of participants with dose reductions | through study completion an average of 6 months
Number of participants with dose interruptions | through study completion an average of 6 months
Dose intensity | through study completion an average of 6 months

SECONDARY OUTCOMES:
The pharmacokinetic (PK) profile of S65487: Area Under the Curve (AUC) | Cycle 1 Day 1, Cycle 1 Day 2, Cycle 1 Day 3 (alternative schedule only), Cyle 1 Day 5 (alternative schedule only), Cycle 1 Day 8, Cycle 1 Day 9, Day 1 of next cycles (one cycle is 21 days)
PK profile of S65487: Volume of distribution at steady-state (Vss) | Cycle 1 Day 1, Cycle 1 Day 2, Cycle 1 Day 3 (alternative schedule only), Cyle 1 Day 5 (alternative schedule only), Cycle 1 Day 8, Cycle 1 Day 9, Day 1 of next cycles (one cycle is 21 days)
PK profile of S65487: total CLearance (CL) | Cycle 1 Day 1, Cycle 1 Day 2, Cycle 1 Day 3 (alternative schedule only), Cyle 1 Day 5 (alternative schedule only), Cycle 1 Day 8, Cycle 1 Day 9, Day 1 of next cycles (one cycle is 21 days)
PK profile of S65487: terminal half-life (t½z) | Cycle 1 Day 1, Cycle 1 Day 2, Cycle 1 Day 3 (alternative schedule only), Cyle 1 Day 5 (alternative schedule only), Cycle 1 Day 8, Cycle 1 Day 9, Day 1 of next cycles (one cycle is 21 days)
Best Overall Response (BOR) | Through study completion, an average of 6 months
  Best Response observed during the treatment period
Overall Response Rate (ORR) | Through study completion, an average of 6 months
  Proportion of patients in whom a complete response (CR) or a partial response (PR)

CONTACTS AND LOCATIONS:
Locations (11):
- The Alfred Hospital Malignant Haematology & Stem Cell Transplantation Services, Melbourne, Victoria, Australia
- France (3):
  - Centre Hospitalier Universitaire Régionale de Lille Hôpital Huriez, Lille
  - CHU Nantes Hôtel Dieu, Nantes
  - CHU de Nice - Hôpital l'Archet 1 Hématologie clinique, Nice
- Spain (4):
  - Clinica Universidad de Navarra, Madrid
  - Clínica Universidad Navarra- Servicio de Hematología, Pamplona
  - Hospital Clínico Universitario de Salamanca- Servicio de Hematología (4a planta), Salamanca
  - Hospital Universitario La Fe - Servicio de Hematología - Torre F - Planta 7, Valencia
- United Kingdom (3):
  - King's College Hospital NHS Foundation Trust, London
  - The Christie NHS foundation Trust, Manchester
  - Freeman Hospital, Newcastle

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: https://clinicaltrials.servier.com/

REFERENCES:
- See also: Find Results on Servier Clinical Trial Data website — https://clinicaltrials.servier.com/
- Available data/document: Individual Participant Data Set — https://clinicaltrials.servier.com/
- Available data/document: Study Protocol — https://clinicaltrials.servier.com/
- Available data/document: Statistical Analysis Plan — https://clinicaltrials.servier.com/
- Available data/document: Informed Consent Form — https://clinicaltrials.servier.com/
- Available data/document: Clinical Study Report — https://clinicaltrials.servier.com/
- Available data/document: Study-level clinical trial data — https://clinicaltrials.servier.com/